CLINICAL TRIAL: NCT06883448
Title: The SUITS Study: Implementation of Home Monitoring in Patients With Pulmonary Fibrosis
Brief Title: Implementation of Home Monitoring in Patients With Pulmonary Fibrosis
Acronym: SUITS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Zuyderland Medisch Centrum, Sittard-Geleen, the Netherlands (Unknown); Leiden University Medical Center, LUMC, Leiden, The Netherlands (Unknown); UMC Utrecht, Utrecht, the Netherlands (Unknown); Rijnstate, Arnhem, the Netherlands (Unknown); Catharina, Eindhoven, the Netherlands (Unknown); MC Leeuwarden, Leeuwarden, the Netherlands (Unknown); OLVG, Amsterdam, the Netherlands (Unknown); Medical Center Haaglanden, The Hague, The Netherlands (Unknown); Amphia, Breda, the Netherlands (Unknown); St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Marlies Wijsenbeek, Prof. Dr., MD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MEC-2024-0045; 10140292110006 (Other Grant/Funding Number: The Netherlands Organisation for Health Research and Development (ZonMw))
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Fibrosis; Interstitial Lung Disease (ILD)
Keywords: eHealth; Hybrid care; Self-management
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned in a 1:1 ratio to receive either hospital-based care or the home monitoring program integrated into hospital-based care. Randomisation will be done with a computer-generated schedule (ALEA Screening and Enrolment Application Software), using block-randomisation, stratified for study site and use of anti-fibrotic treatment (yes or no).
Masking Description: Participants, health-care providers, and research staff will not be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital-based care (No Intervention): Hospital-based care involves outpatient clinic visits every three months including in-hospital lung function testing.
- Home monitoring care (Experimental): Patients in the home monitoring group will receive a home spirometer, pulse oximetry meter, and access to a smartphone or tablet app, where they can perform home based measurements weekly and complete PROMs. Furthermore, this app includes disease specific information and allows for direct communication with the hospital via eConsultation. In the home monitoring group, half of the outpatient clinic visits will alternately be replaced by remote visits via video consultation.
  Interventions: Combination Product: Home monitoring care

INTERVENTIONS:
Combination Product: Home monitoring care — Patients in the home monitoring group will receive a home spirometer, pulse oximetry meter, and access to a smartphone or tablet app, where they can perform home based measurements weekly and complete PROMs. Furthermore, this app includes disease specific information and allows for direct communication with the hospital via eConsultation. In the home monitoring group, half of the outpatient clinic visits will alternately be replaced by remote visits via video consultation.
  Arms: Home monitoring care

SUMMARY:
The objective of this study is to evaluate the impact of structurally replacing half of the outpatient clinic visits for patients with pulmonary fibrosis by home monitoring and video consultations on patient self-management and health(care) outcomes.

DETAILED DESCRIPTION:
Patients will be randomly assigned to receive either hospital-based care or a home monitoring program integrated into hospital-based care. Hospital-based care involves outpatient clinic visits every three months including lung function testing. Home monitoring involves weekly measurements of both physiological- and patient reported outcomes (PROs) in a mobile health care application with half of the outpatient clinic visits alternately being replaced by remote video consultations. The home monitoring program includes home spirometry, pulse-oximetry, PROs, video consultations, a medication coach, and an infotheque showing disease-specific information. Questionnaires will be filled out by both study groups at set time points. The total study duration for individual patients will be 12 months.

Trial Registration and Ethics Statement In the Netherlands, clinical trial registration is not mandatory for studies exempt from ethics review. As this study was exempt from ethics review, as approved by the IRB of Erasmus Medical Center in Rotterdam, the Netherlands, the study was not prospectively registered. During the enrollment phase, the study protocol was retrospectively registered on ClinicalTrials.gov to ensure public access to the study protocol and study outcomes. IRB approval was obtained prior to enrollment of the first participant. No changes were made to the IRB-approved study protocol (version 1, 11-01-2024) prior to registration on ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* A multidisciplinary ILD team diagnosis of pulmonary fibrosis according to ATS/ERS/JRS/ALAT guidelines;
* Adults (=/>18 years).

Exclusion Criteria:

* Patients who are not able to speak, read and/or write in Dutch;
* Patients with no access to the internet;
* Patients with a life expectancy of less than 1 year as determined by the treating healthcare provider;
* Patients who are or have been using a home monitoring program for PF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient self-management | Baseline to 12 months
  Delta score of the Patient Activation Measure (PAM) questionnaire. The PAM is a 13-item survey assessing levels of patient activation in terms of managing their own health and healthcare. Total score ranges are 0-100, with higher scores indicating greater patient activation.

SECONDARY OUTCOMES:
Patient self-management | Baseline
  The Patient Activation Measure (PAM) questionnaire is a 13-item survey assessing levels of patient activation in terms of managing their own health and healthcare. Total score ranges are 0-100, with higher scores indicating greater patient activation.
Patient self-management | Baseline to 6 months
  Delta score of the Patient Activation Measure (PAM) questionnaire. The PAM is a 13-item survey assessing levels of patient activation in terms of managing their own health and healthcare. Total score ranges are 0-100, with higher scores indicating greater patient activation.
Living with Pulmonary Fibrosis (L-PF) questionnaire | Baseline
  The Living with Pulmonary Fibrosis (L-PF) questionnaire is developed to assess symptoms and HRQOL in patients with Pulmonary Fibrosis. It consists of 44 items divided into two modules: symptoms (23 items) and impacts (21 items). The symptom module assesses shortness of breath, cough and fatigue. The impacts module assesses multiple aspects of HRQOL on a five-option numeric rating score. Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.
Living with Pulmonary Fibrosis (L-PF) questionnaire | Baseline to 6 months
  Delta scores of all domains of the Living with Pulmonary Fibrosis (L-PF) questionnaire will be assessed. The L-PF questionnaire is developed to assess symptoms and HRQOL in patients with Pulmonary Fibrosis. It consists of 44 items divided into two modules: symptoms (23 items) and impacts (21 items). The symptom module assesses shortness of breath, cough and fatigue. The impacts module assesses multiple aspects of HRQOL on a five-option numeric rating score. Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.
Living with Pulmonary Fibrosis (L-PF) questionnaire | Baseline to 12 months
  Delta scores of all domains of the Living with Pulmonary Fibrosis (L-PF) questionnaire will be assessed. The L-PF questionnaire is developed to assess symptoms and HRQOL in patients with Pulmonary Fibrosis. It consists of 44 items divided into two modules: symptoms (23 items) and impacts (21 items). The symptom module assesses shortness of breath, cough and fatigue. The impacts module assesses multiple aspects of HRQOL on a five-option numeric rating score. Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.
King's brief Interstitial Lung Disease Health Status (K-BILD) | Baseline
  The K-BILD health status questionnaire is a 15-item validated, self-completed heath status questionnaire. It contains three domains: breathlessness and activities, psychological and chest symptoms. The total score ranges are 0-100, with higher scores corresponding with better HRQOL.
King's brief Interstitial Lung Disease Health Status (K-BILD) | Baseline to 6 months
  Delta scores of all domains of the King's brief Interstitial Lung Disease Health Status (K-BILD) questionnaire will be assessed. The K-BILD health status questionnaire is a 15-item validated, self-completed heath status questionnaire. It contains three domains: breathlessness and activities, psychological and chest symptoms. The total score ranges are 0-100, with higher scores corresponding with better HRQOL.
King's brief Interstitial Lung Disease Health Status (K-BILD) | Baseline to 12 months
  Delta scores of all domains of the King's brief Interstitial Lung Disease Health Status (K-BILD) questionnaire will be assessed. The K-BILD health status questionnaire is a 15-item validated, self-completed heath status questionnaire. It contains three domains: breathlessness and activities, psychological and chest symptoms. The total score ranges are 0-100, with higher scores corresponding with better HRQOL.
The EuroQol five dimensions 5-level plus respiratory bolt-on (EQ-5D-5L+R) questionnaire | Baseline
  The EQ-5D-5L+R questionnaire is a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises six dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and respiratory complaints on a 5-point scale. From these 6 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better quality of life.
The EuroQol five dimensions 5-level plus respiratory bolt-on (EQ-5D-5L+R) questionnaire | Baseline to 6 months
  Delta scores of the EuroQol five dimensions 5-level plus respiratory bolt-on (EQ-5D-5L+R) questionnaire will be assessed. The EQ-5D-5L+R questionnaire is a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises six dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and respiratory complaints on a 5-point scale. From these 6 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better quality of life.
The EuroQol five dimensions 5-level plus respiratory bolt-on (EQ-5D-5L+R) questionnaire | Baseline to 12 months
  Delta scores of all dimensions of the The EuroQol five dimensions 5-level plus respiratory bolt-on (EQ-5D-5L+R) questionnaire will be assessed. The EQ-5D-5L+R questionnaire is a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises six dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and respiratory complaints on a 5-point scale. From these 6 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better quality of life.
Scheduled respiratory related outpatient clinic visits | Baseline to 12 months
Unscheduled respiratory related outpatient clinic visits | Baseline to 12 months
Respiratory related remote consultations | Baseline to 12 months
  Compare the number of remote consultations performed.
Respiratory related emergency visits | Baseline to 12 months
Respiratory related hospitalisations | From baseline to 12 months
Mortality or lung transplantation | Baseline to 12 months
Forced vital capacity (FVC) | Baseline
  Forced vital capacity (FVC) measured with pulmonary function study (PFT) as ml and as percentage predicted of healthy standards (in %).
Forced vital capacity (FVC) | Baseline to 6 months
  Delta forced vital capacity (FVC) measured with pulmonary function study (PFT) as ml and as percentage predicted of healthy standards (in %).
Forced vital capacity (FVC) | Baseline to 12 months
  Delta forced vital capacity (FVC) measured with pulmonary function study (PFT) as ml and as percentage predicted of healthy standards (in %).
Diffusing capacity of the lung for carbon monoxide (DLCO) | Baseline
  Diffusing capacity of the lungs for carbon monoxide (DLCO) measured with pulmonary function study (PFT) as ml and as percentage predicted of healthy standards (in %).
Diffusing capacity of the lung for carbon monoxide (DLCO) | Baseline to 6 months
  Delta diffusing capacity of the lungs for carbon monoxide (DLCO) measured with pulmonary function study (PFT) as ml and as percentage predicted of healthy standards (in %).
Diffusing capacity of the lung for carbon monoxide (DLCO) | Baseline to 12 months
  Delta diffusing capacity of the lungs for carbon monoxide (DLCO) measured with pulmonary function study (PFT) as ml and as percentage predicted of healthy standards (in %).
Forced vital capacity (FVC) | Baseline
  Forced vital capacity (FVC) measured with home measured pulmonary function study (PFT) as ml and as percentage predicted of healthy standards (in %).
Forced vital capacity (FVC) | Baseline to 6 months
  Delta forced vital capacity (FVC) measured with home measured pulmonary function study (PFT) as ml and as percentage predicted of healthy standards (in %).
Forced vital capacity (FVC) | Baseline to 12 months
  Delta forced vital capacity (FVC) measured with home measured pulmonary function study (PFT) as ml and as percentage predicted of healthy standards (in %).
Correlation and agreement of home measured Forced vital capacity (FVC) | From baseline to 12 months
  Correlations between home measured Forced vital capacity (FVC) and in-hospital FVC in ml in the home monitoring group.
Patient adherence to home monitoring protocol | Baseline to 12 months
  Patients' adherence to home monitoring for home measured spirometry, pulse-oximetry, and patient-reported outcome measures (PROMs).

OTHER OUTCOMES:
Cost-effectiveness and cost-utility analyses | Baseline to 12 months
  The costs, cost-effectiveness and cost-utility analyses will be conducted from a healthcare system and societal perspective.
Healthcare professional- and patient satisfaction | 12 months
  Healthcare providers and patients will be asked about their satisfaction and experiences on home monitoring.
Time to detection of a decline of 10% in in-hospital versus home-based FVC | Baseline to 12 months
Travel movements | Baseline to 12 months
  Explorative evaluation of the effect of home monitoring on travel movements.

CONTACTS AND LOCATIONS:
Overall Officials: Marlies S. Wijsenbeek-Lourens, Prof Dr, Principal Investigator — Department of Respiratory Medicine, Center of Excellence for Interstitial Lung Disease, Erasmus University Medical Center, Rotterdam, The Netherlands
Locations (11):
- Netherlands (11):
  - Department of Pulmonology, Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Department of Pulmonary Diseases, Rijnstate Hospital, Arnhem
  - Department of Respiratory Medicine, Amphia Hospital, Breda
  - Department of Respiratory Medicine, Catharina Hospital, Eindhoven
  - Department of Pulmonary Medicine, Zuyderland Medical Centre, Heerlen
  - Department of Pulmonology, Medical Center Leeuwarden, Leeuwarden
  - Department of Pulmonology, Leiden University Medical Center, Leiden
  - Interstitial Lung Diseases Center of Excellence, Department of Pulmonology, St Antonius Hospital, Nieuwegein
  - Department of Respiratory Medicine, Center of Excellence for Interstitial Lung Disease, Erasmus University Medical Center, Rotterdam
  - Department of Pulmonology, Haaglanden Medisch Centrum, The Hague
  - Division of Heart and Lungs, University Medical Center Utrecht and Utrecht University, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided